CLINICAL TRIAL: NCT02952326
Title: Comparison Of The Effect of Adding XP Endo Finisher To The Irrigation Protocol Versus Conventional Irrigation Method On Post-Operative Flare Ups In Necrotic Teeth
Brief Title: Comparing Between XP Endo Finisher and Conventional Irrigation Method On Post-Operative Flare Ups In Necrotic Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghada Ihab Mohamed, Resident at Endodontic department, faculty of oral and dental medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XP and Protaper next
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Dental Pulp Necroses
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- XP Endo Finisher (Experimental)
  Interventions: Procedure: XP Endo Finsher as final step of the irrigation protocol
- Conventional needle irrigation (Active Comparator)
  Interventions: Procedure: Conventional needle irrigation only

INTERVENTIONS:
Procedure: XP Endo Finsher as final step of the irrigation protocol — The canals will be thoroughly irrigated using 3ml syringe of 2.5% Sodium hypochlorite between every subsequent instrument. XP Endo finisher is used after the last instrument in preparation
  Arms: XP Endo Finisher
Procedure: Conventional needle irrigation only — The canals will be thoroughly irrigated using 3ml syringe of 2.5% Sodium hypochlorite between every subsequent instrument.
  Arms: Conventional needle irrigation

SUMMARY:
Comparing the postoperative flare ups and pain after adding the XP Endo Finisher to the final irrigation protocol on necrotic mandibular premolars.

DETAILED DESCRIPTION:
patients are randomized into 2 groups after meeting the eligibility criteria,

1. Each patient will be given pain scale chart in order to record his /her pain level before any intervention.
2. The tooth is anesthetized, accessed and mechanical instrumentation to be made 3 A) For the experimental group: The canals will be thoroughly irrigated using 3ml syringe of 2.5% Sodium hypochlorite between every subsequent instrument. XP Endo finisher is used after the last instrument in preparation

B) For the control group :

The canals will be thoroughly irrigated using 3ml syringe of 2.5% Sodium hypochlorite between every subsequent instrument.

4) Obturation is done and postoperative instructions are given to the patient

ELIGIBILITY:
Inclusion Criteria:

i. Age between 18-50 years old. ii. Males or Females. iii. mandibular Premolars

* Asymptomatic.
* Non-vital response of pulp tissue (negative response).
* With or without periapical radiolucency.

Exclusion Criteria:

i. Patients allergic to penicillin. ii. Pregnant females. iii. Patients having significant systemic disorder. iv. If antibiotics have been administrated during the past two weeks preoperatively.

v. Patients having bruxism or clenching. vi. Teeth that have :

* Vital pulp tissues.
* Association with swelling
* Acute peri-apical abscess
* Periodontally affected teeth
* No possible restorability
* Previous endodontic treatment.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-11 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain recorded by the patient using a four step pain scale (0-3) | up to 5 days after the treatment

SECONDARY OUTCOMES:
Post-operative swelling | up to 5 days after the treatment
Need\ number of Analgesic tablets | up to 5 days after the treatment
Need for systemic antibiotics | up to 5 days after the treatment

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elnaghy AM, Mandorah A, Elsaka SE. Effectiveness of XP-endo Finisher, EndoActivator, and File agitation on debris and smear layer removal in curved root canals: a comparative study. Odontology. 2017 Apr;105(2):178-183. doi: 10.1007/s10266-016-0251-8. Epub 2016 May 20. PMID 27206916
- [Background] Siqueira JF Jr. Microbial causes of endodontic flare-ups. Int Endod J. 2003 Jul;36(7):453-63. doi: 10.1046/j.1365-2591.2003.00671.x. PMID 12823700